CLINICAL TRIAL: NCT01073995
Title: The Effectiveness of Selective Nerve Root Injections in Preventing the Need for Surgery in Patients With Lumbar Disc Herniations
Brief Title: The Effectiveness of Selective Nerve Root Injections in Preventing the Need for Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Dr. neil Manson, Orthopaedic surgeon, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-1376
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Radiculopathy
Keywords: Radiculopathy; Sciatica; Lumbar Disc Herniation; Surgical Alternative
MeSH Terms: conditions — Radiculopathy; Sciatica; Intervertebral Disc Displacement | interventions — Triamcinolone Acetonide; Bupivacaine; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kenalog and Sensorcaine (Active Comparator): The following drugs will be administered during a one time injection of the appropriate spinal level based off clinical and radiographic information:
  Intervention:
  Kenalog 40 mg/ml and Sensorcaine 0.25% 1cc
  Interventions: Drug: Kenalog and Sensorcaine
- Saline (Placebo Comparator): Saline injections will be used to mimic the Steroid dose
  Interventions: Drug: Kenalog and Sensorcaine

INTERVENTIONS:
Drug: Kenalog and Sensorcaine — Kenalog: 40 mg/ml Sensorcaine 0.25%: 1cc
  Other Names: Kenalog; Triamcinolone; Sensorcaine; Marcaine; Bupivacaine hydrochloride

SUMMARY:
The median Orthopaedic surgery wait time in Canada is 36.7 weeks (Esmail 2008), thus there is a need to find alternative treatments for pathologies such as lumbar disc herniations (LDH). The literature has demonstrated that selective nerve root injections (SNRI) are able to alleviate sciatic symptoms caused by LDH (Riew 2006) and may be beneficial as an alternative to surgery. It is necessary to determine whether SNRIs provide significant symptom resolution alleviating the need for surgery, or to determine if their success is transient and delays the time to surgery. The purpose of the proposed study is to evaluate the success of SNRI in patients suffering with LDH and to determine which factors influence outcome. Over the span of 2 years, data from 100 patients will be collected. These patients will be surgical candidates and have exhausted all non-operative measures prior to receiving a SNRI. Upon first assessment, each eligible patient will be randomly assigned to the treatment (steroid) or control (saline) group. The patient and all treating physicians will be blinded to the treatment given. Each patient will be followed over their course of treatment and information pertaining to their pain and symptoms will be recorded using standard questionnaires. Patient demographics, diagnosis, Worker's Compensation status, spinal levels treatment/outcome, and time from referral to treatment will also be evaluated. The primary outcome measure will be defined as the avoidance of surgery.

DETAILED DESCRIPTION:
Patient Selection: All patients (ages 18-65 years) who have been diagnosed with lower extremity radiculopathy (sciatica) secondary to a lumbar disc herniation that have been referred for SNRI by the principal investigator (Dr. Neil Manson) will be asked to participate in the study. All patients will have exhausted non-operative measures.

Initial Assessment: During the initial office visit, patients will be assessed by the principle investigator for inclusion in the study. If the patient demonstrates interest in the proposed research they will be provided a Consent Form and given the opportunity to ask a Research Assistant questions regarding their participation.

. Injections: Standard procedures for SNRI will be used by the participating Radiologists in the Department of Radiology at the Saint John Regional Hospital. Each patient will be randomly assigned by a Research Assistant to either the treatment (Kenalog/Sensorcaine) or control (Saline) group. All treatments will be blinded to the treating physicians and the patient.

Injectates: Control Group: Saline Treatment Group: Kenalog 40cc/0.25% Sensorcaine

Follow up assessment: During a follow-up visit, patients will be re-assessed to determine the success of the injection. SNRI success will be determined by self-reported pain and symptom reduction. If the patient and principle investigator do not deem the injection successful, further treatment options will be discussed (second injection, surgery, etc) and follow-up evaluations will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* Diagnosed with lower extremity radiculopathy (sciatica) secondary to a lumbar disc herniation
* Exhausted non-operative measures:
* Medication has not been helpful in treating the patient's pain/symptoms
* Modification of daily activities has not been helpful in treating the patient's pain/symptoms
* Physiotherapy has not been helpful in treating the patient's pain/symptoms.
* Patient of the Investigator
* Patient willing to proceed with surgical intervention

Exclusion Criteria:

* Age: < 18 or > 65
* Any patient who has not attempted conservative non-operative treatment for a minimum of 6 weeks
* Any patient who has not been deemed a surgical candidate
* Any patient who has a contraindication for surgery
* Any patient who has a contraindication for Kenalog or Sensorcaine
* Known sensitivity to medicinal or non-medicinal ingredients
* Systemic infection
* Idiopathic thrombocytopenic purpura
* Cerebrospinal diseases
* Pregnancy and nursing mothers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Surgical Avoidance | 5 years
  After a minimum 1 year follow-up of an SNRI, a statistical analysis will be conducted to determine group differences in surgical necessity

SECONDARY OUTCOMES:
Subjective questionnaires | 5 Years
  Each patient will be followed over their course of treatment and information pertaining to their pain and symptoms will be recorded using standard questionnaires such as the SF-36 Questionnaire, the Oswestry Disability Index, and the Visual Analogue Scale. Patient demographics, diagnosis, Worker's Compensation status, spinal levels treatment/outcome, and time from referral to treatment will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Manson, MD, Principal Investigator — Canada East Spine Centre; Erin E Bigney, MA, Study Director — Canada East Spine Center
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Yes
Manuscript preparation in progress